CLINICAL TRIAL: NCT03096132
Title: Effect of Treatment Dose on Childhood Obesity
Brief Title: FRESH-DOSE: Families Responsibility Education Support Health-Dual Options for Sustained Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160289; R01DK108686 (NIH)
Record Dates: First submitted 2017-03-09; First posted 2017-03-30 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Overweight; Obesity
Keywords: Obesity; Overweight; Overeating; Body Mass Index; Treatment; Intervention; Family Based Therapy; Weight; Children
MeSH Terms: conditions — Overweight; Obesity; Hyperphagia; Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Based Behavioral Treatment (Active Comparator): The program includes information about diet and physical activity education, in addition to parent management skills and behavior therapy strategies in a weekly group setting.
  Interventions: Behavioral: Family Based Behavioral Treatment
- Guided Self-Help Fam. Based Bx Treatment (Experimental): The program includes information about diet and physical activity education, in addition to parent management skills and behavior therapy strategies in a guided self-help manual.
  Interventions: Behavioral: Guided Self-Help Fam. Based Bx Treatment

INTERVENTIONS:
Behavioral: Family Based Behavioral Treatment — Treatment includes 20 90 minute visits over 6 months which include 60 min parent and child separate groups and 30 min behavioral coaching. FBT includes information regarding nutrition and physical activity, as well as behavior therapy skills, including parenting skills, self-monitoring, problem solving skills, motivation systems, emotional regulation, stress management, stimulus control, and relapse prevention.
  Other Names: FBT
  Arms: Family Based Behavioral Treatment
Behavioral: Guided Self-Help Fam. Based Bx Treatment — Treatment includes 14 20 minute visits over 6 months. gshFBT is delivered to parent/child dyads and includes the same content in the FBT groups but it is provided in a manual. The 20-minute visits focus on clarifying information in the manuals, collecting weight and self-monitoring logs, and problem solving any barriers to implementation.
  Other Names: gshFBT
  Arms: Guided Self-Help Fam. Based Bx Treatment

SUMMARY:
The objective of the study is to evaluate whether a less intensive intervention, Guided Self-Help Family Based Treatment (gshFBT), is non-inferior to the more intensive Family Based Treatment (FBT) for childhood obesity on child weight loss over 18-months. Cost-effectiveness of both treatments will also be compared.

DETAILED DESCRIPTION:
The primary aim of this project is to determine whether gshFBT is non-inferior to FBT for childhood obesity on child weight loss. Four assessments will be conducted; baseline (month 0), month 6 (post-treatment), and at month 12 and month 18. Assessments will include the following for child and parent: anthropometry, physical activity, nutrition, and cost-effectiveness. Cost-effectiveness will be calculated from a societal perspective and a third party payor perspective. This program of research has the potential to advance the standard of practice for children who are overweight or obese by providing a less intensive but more cost-effective intervention.

ELIGIBILITY:
1. An overweight child age 7-12, whose BMI is ≥ 85th percentile but does not meet criteria for severe obesity (i.e., BMI ≥120% of the 95th percentile or an absolute BMI ≥ 35 kg/m2 , whichever is lower for age and gender)
2. The parent willing to participate can read English at a minimum of a 5th grade level
3. Parent and Child willing to commit to attending all treatment and assessment sessions and be randomized to either treatment arm
4. Child or parent is free from psychiatric illness than may affect participation;
5. Child does not have any medical conditions that impact weight or may affect participation in physical activity or treatment
6. Child is not taking medications that may impact their weight (unless medication dosage is stable and not for the purpose of impacting weight and appetite)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Child weight loss | Change from baseline to month 6, 12 and 18
  BMI; BMIz
Cost-effectiveness | Baseline to month 6, 12 and 18
  Cost per .1 BMIz change in child weight including health care costs, participant costs and treatment costs.

SECONDARY OUTCOMES:
Parent BMI | Change from baseline to month 6, 12 and 18
  BMI
Child Physical Activity - minutes of moderate-vigorous activity | Change from baseline to month 6, 12 and 18
  Measured by accelerometer, minutes in Moderate to Vigorous physical activity
Parent Physical Activity - minutes of moderate-vigorous activity | Change from baseline to month 6, 12 and 18
  Measured by accelerometer, minutes in Moderate to Vigorous physical activity
Child Nutrition-measured as servings of fruit and vegetables per day | Change from baseline to month 6, 12 and 18
  Self-reported number of servings of fruits and vegetables consumed each day
Parent Nutrition-measured as servings of fruit and vegetables per day | Change from baseline to month 6, 12 and 18
  Self-reported number of servings of fruits and vegetables consumed each day

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States

REFERENCES:
- [Background] Accurso EC, Norman GJ, Crow SJ, Rock CL, Boutelle KN. The role of motivation in family-based guided self-help treatment for pediatric obesity. Child Obes. 2014 Oct;10(5):392-9. doi: 10.1089/chi.2014.0023. Epub 2014 Sep 2. PMID 25181608
- [Background] Boutelle KN, Norman GJ, Rock CL, Rhee KE, Crow SJ. Guided self-help for the treatment of pediatric obesity. Pediatrics. 2013 May;131(5):e1435-42. doi: 10.1542/peds.2012-2204. Epub 2013 Apr 1. PMID 23545372